CLINICAL TRIAL: NCT07381894
Title: Multicentre Hypertrophic Cardiomyopathy Registry
Status: Not yet recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Wei Jun How, Cardiologist, University of Manchester
Other Study IDs: 363346
Record Dates: First submitted 2025-12-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common inherited heart condition, affecting approximately 1 in 500 people. It causes the heart muscle to thicken, which can lead to blockages in blood flow (left ventricular outflow tract obstruction), shortness of breath, and an increased risk of heart failure or sudden cardiac arrest.

While standard treatments exist and new targeted medications (cardiac myosin inhibitors) have recently been approved, doctors still need better data to predict which treatments will work best for each individual patient. This national registry based in the UK is a secure database that collects health information from HCM patients across multiple NHS hospital sites in the UK over several years.

Participants in this study will have their routine health information collected from their medical records, including details from heart scans (echocardiograms and MRIs), blood tests, and genetic information. With this HCM registry, we aim to improve disease understanding and risk prediction, paving the way for more personalised treatment plans for the HCM community in the future

DETAILED DESCRIPTION:
Study Overview:

The National Hypertrophic Cardiomyopathy (HCM) Registry is a prospective, multicentre, observational registry designed to characterize contemporary UK clinical practice and provide longitudinal, granular phenotyping of patients with HCM. The study aims to recruit approximately 2,500 participants across multiple NHS hospitals over a 5-year enrollment period.

Primary Objectives:

Describe the natural history and treatment response of HCM across UK centers, including the utilisation and outcomes of medical therapies, including cardiac myosin inhibitors (CMIs).

Secondary Objectives:

Determine the incidence and predictors of clinically significant arrhythmias. Define genotype-phenotype correlations. Correlate serum biomarkers (e.g., NT-proBNP, high-sensitivity cardiac troponin) and multimodality imaging metrics (echocardiographic strain, CMR-derived scar burden) with clinical outcomes.

Study Population and Procedures:

Eligible participants include adults (above the age of 18 years old) with a definite clinical diagnosis of HCM, not explained by abnormal loading conditions.

Data collection occurs during routine clinical visits with collected variables including demographics, comorbidities, medications, 12-lead ECG, biomarkers, echocardiography, CMR parameters, and device status (if available). All clinical care remains at the discretion of the treating physician.

Data Management: Participants are pseudonymized with a unique study ID and entered into a secure database.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Hypertrophic Cardiomyopathy (HCM) clinically and not solely explained by abnormal loading conditions (e.g., significant hypertension, valvular disease

Exclusion Criteria:

* Participants who do not fulfil the imaging and clinical diagnostic criteria of HCM

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of hypertrophic cardiomyopathy will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Key Efficacy Parameters (LVOT Gradient) | 3-5 years
  Change in left ventricular outflow tract (LVOT) gradient (measured echocardiographically in mmHg) at both resting and stress condition in obstructive cases in response to treatment

SECONDARY OUTCOMES:
Incidence of Clinically Significant Arrhythmias | 5 years
  Incidence rates of new-onset or recurrent atrial fibrillation (AF)/atrial flutter (AFL) and sustained/non-sustained ventricular tachycardia (VT/NSVT) episodes.
Correlation of Genotype and Imaging with Clinical Outcomes | 5 years
  Correlation analysis to define genotype-phenotype relationships, and the relationship between imaging-derived parameters such as scar burden (Late Gadolinium Enhancement, LGE) and clinical outcomes.
Change in Serum Biomarker | 3-5 years
  Response in cardiac biomarker profile (nT-proBNP measured in ng/L and serum troponin measured in ng/L) in response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided